CLINICAL TRIAL: NCT00653172
Title: A Double-Blind, Multicenter, Randomized, Double Dummy, Three-Arm Parallel-Group Comparative Study of the Efficacy, Safety and Tolerance of Oral NXL 103 Versus Oral Comparator in the Treatment of Community-Acquired Pneumonia in Adults
Brief Title: Comparative Study of NXL103 Versus Comparator in Adults With Community Acquired Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novexel Inc (Industry)
Responsible Party: Dr. Carole A. Sable Chief Medical Officer, Novexel SA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NXL103/2001
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Community Acquired Pneumonia
Keywords: CAP; community acquired pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — flopristin, linopristin drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): NXL103
  Interventions: Drug: NXL103
- 3 (Active Comparator)
  Interventions: Drug: comparator
- 2 (Experimental): NXL103
  Interventions: Drug: NXL103

INTERVENTIONS:
Drug: NXL103 — 600mg orally twice daily
  Arms: 2
Drug: comparator — comparator twice daily
  Arms: 3
Drug: NXL103 — 500mg orally twice daily
  Arms: 1

SUMMARY:
The purpose of this study is to compare the efficacy, safety and tolerance of 2 different dose levels of oral NXL103 with oral comparator in the treatment of community acquired pneumonia in adults

ELIGIBILITY:
Inclusion Criteria:

* Community acquired pneumonia

Exclusion Criteria:

* severe CAP
* respiratory infections attributed to sources other than community acquired bacterial infection
* concomitant pulmonary disease
* history of hypersensitivity to study medication, macrolide or beta lactam antibiotics

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Evaluate Clinical outcome | early follow up visit (day 14 to 21)

SECONDARY OUTCOMES:
Evaluate bacteriological outcome | early follow up visit (day 14 to 21)
Evaluate safety | first dose, throughout treatment, and to follow up visit

CONTACTS AND LOCATIONS:
Locations (60):
- Chile (4):
  - Clinica de Enfermedades Resp. "Miguel de Servet" SA, Santiago
  - Complejo Asistencial Barros Luco Trudeau, Santiago
  - Hospital de Urgencia Asistencia Publica, Santiago
  - Hospital Regional de Rancagua, Santiago
- Croatia (3):
  - Clinic for infectious diseases, Zagreb
  - General Hospital Sveti Duh, Zagreb
  - University Hospital Dubrava, Zagreb
- Estonia (5):
  - Linnamoisa Perearstikeskus, Tallinn
  - Merelahe Family Doctors Centre, Tallinn
  - Nolvaku Family Doctor Center, Tartu
  - Pullerits & Peda Perearstikeskus, Tartu
  - Marje Toom Family Doctors Practice, Võru
- Germany (5):
  - Penumologen=Praxis Lichterfelde, Berlin
  - Asklepios Klinik St. Georg, Hamburg
  - Asklepiosklinik Wandsbeck, Hamburg
  - Praxis Dr. H. Mueller, Potsdam
  - Praxis Dr. W. Wyborski, Werneck
- Peru (2):
  - Hospital Nacional Arzobispo Loayza, Lima
  - Hospital Nacional Guillermo Almenara, Lima
- Poland (10):
  - Indywidualna Specjalistyczna Praktyka Lekarska, Bialystok
  - SP ZOZ Wojewodzki Szpital Specjalistyczny im., Bialystok
  - SPZOZ Osrodek Zdrowia wBienkowce, Bieńkowice
  - NZOZ Poradnia Medycyny Rodzinnej, Gdansk
  - Nzoz "Esculap", Gniewkowo
  - Prywatny Gabinet Specjalistyczny, Lodz
  - SP ZOZ Wielkopolskie Centrum Chrob, Poznan
  - Nzoz "Mig'Med", Wąbrzeźno
  - NZOZ Centrum Badan Klinicznych, Wroclaw
  - Wojewodzki Szpital we wloclawku, Włocławek
- Romania (9):
  - Spitalul Clinical Judetean de Urgenta, Brasov
  - Centrul de Diagnostic si Tratament "Dr. Victor Babes", Bucharest
  - Spitalul Clinic de Urgenta Bucuresti, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Spitalul Universitar de Urgenta Elias, Bucharest
  - Dispensarul TB nr. 1 Galati, Galati
  - Spitalul de Pneumologie Galati, Galati
  - Spitalul Judetean de Urgenta "Sf. loan cel, Suceava
  - Centrul Medical Privat "Medicali's", Timosoara
- South Africa (13):
  - Langeberg Medical Centre, Cape
  - GCT Trial Centre, Mercantile Hospital, E Cape
  - Rabie, W, Free State
  - Rubins Building, Free State
  - Benmed Park Clinical, Gauteng
  - Clinresco Centres (Pty) Ltd, Gauteng
  - DJW Navorsing, Gauteng
  - Eastmed Medical Centre, Gauteng
  - Intercare-Medical & Dental Centre, Gauteng
  - Jubilee Hospital, Gauteng
  - Sebastian, P, KZ-Natal
  - Pretoria West Medicross, Pretoria West
  - Clinical Project Research, Worcester
- Ukraine (9):
  - DSMA b. on Dnepropetrovsk City Clin. Hosp. #6, Dnipro
  - DSMU n.a. M. Gorkyy, Don.Reg.Territorial Med. Clin Ass., Donetsk
  - Iv-Frank St. Med Uni. b.o.lv Frank. Centr City Clin. Hospital, Frankovsk
  - Kharkiv City Clinical Hospital # 13, Kharkiv
  - City Tuberculosis Hospital # 1, Kiev
  - F.G. Yanovskyy Inst. of Ph. & Pulm. of Ac. of Med. Scien. of Ukr, Kiev
  - F.G. Yanovskyy Institute of P & P AMS of Ukr, Kyiv
  - Institute of Therapy AMS Ukr. n.a. Malaya, Mykolayiv
  - Nikolaev City Clinical Hospital # 1, Mykolayiv